CLINICAL TRIAL: NCT05581602
Title: Actimeric Monitoring of the Use of the Paretic Upper Limb in the Activities of Daily Living of the Post-chronic Stroke Subject in a Home Environment
Brief Title: Actimetry Monitoring of the Paretic Upper Limb in Chronic Post Stroke.
Acronym: ParUse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other); IMT Mines Alès (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL21_0512
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Chronic Stroke; Non-use of the Paretic Upper Limb
Keywords: Accelerometry; Stroke; Upper limb; Functional recovery; Home environment; Rehabilitation; Real use; Non use
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The first phase of this project is a bicentric cross-sectional study in 30 hemiparetic post-stroke subjects in chronic phase and 30 healthy subjects, age and gender matched.
  The second phase is a 6-month longitudinal study, in a subgroup of 5 post-stroke subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemiparetic post-stroke subjects (Experimental): Stroke patients with motor sequelae in the upper limb.
  Interventions: Device: Wearing bracelets (3-Axis Logging Accelerometer)
- Healthy subjects (Other): Subjects without stroke.
  Interventions: Device: Wearing bracelets (3-Axis Logging Accelerometer)

INTERVENTIONS:
Device: Wearing bracelets (3-Axis Logging Accelerometer) — Participants will be required to wear wristbands containing an accelerometer on each wrist. The bracelets will be kept on both wrists for 7 days with permission to remove them from time to time.

SUMMARY:
After a stroke, 80% of patients continue to have difficulty using their paretic upper limb in activities of daily living (ADL) despite post-stroke rehabilitation practices that aim to promote the use of the paretic upper limb. It is known that functional recovery depends on actual use (Use it or Loose it), but one-time measurements in the clinic do not allow quantification of the actual use of the paretic upper limb in daily life (in the person's living environment).

The investigators hypothesize the feasibility of quantifying functional use of the paretic upper limb by actimetry in clinical routine.

DETAILED DESCRIPTION:
After a stroke, 80% of patients continue to have difficulty using their paretic upper limb in activities of daily living (ADL) despite post-stroke rehabilitation practices that aim to promote the use of the paretic upper limb. It is known that functional recovery depends on actual use (Use it or Loose it), but one-time measurements in the clinic do not allow quantification of the actual use of the paretic upper limb in daily life (in the person's living environment).

Project will monitor 30 chronic and 30 healthy subjects over one week period using two wrist worn sensors .

The main objective is to objectively quantify by actimetry, over 7 days, the real functional use of the paretic upper limb in the activities of daily living of post-stroke hemiparetic subjects in chronic phase, by the functional use ratio between the two arms (UseRatio).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria common to all participants:

* Be between 18 and 90 years old

Post-stroke subjects should:

* Having a stroke with motor sequelae in the upper limb
* Be in the chronic phase (>3 months post-stroke) of a stroke whatever the aetiology

Exclusion Criteria:

Non inclusion criteria common to all participants:

* Absence of free, informed and express oral consent
* No affiliation to a French social security system or beneficiary of such a system
* Patient protected by law
* Pregnant or breastfeeding women

Not eligible for inclusion, post-stroke subjects:

* Not understanding the constraints of the study
* Have cognitive impairments that prevent them from understanding the study
* With a known hemigligence in the medical record (omission > 8 on bells test)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
FuncUseRatio | 7 days
  The paretic functional use score is a ratio of functional movements performed by the paretic upper limb to the sum of functional movements performed by the paretic and non-paretic upper limbs (in percentage %).

SECONDARY OUTCOMES:
Use | 7 days
  Measurement of the amount of functional movement of each upper limb, in an ecological situation during activities of daily living of post-stroke and healthy subjects.
Intensity | 7 days
  Measurement of the intensity of movements (functional and non-functional) of each upper limb, in an ecological situation during activities of daily living of post-stroke and healthy subjects.
Profil | During intervention
  The activity log is presented in the form of a table. The columns represent the days of recording (Day 1 => Day 7), the rows represent the time slots hour by hour
Motor deficit | During the inclusion visit or information taken in the medical file
  Motor deficit will be measured by the Fugl-Meyer Upper Extremity (FM-UE)
Dispersion of UseRatio | 6 months
  The dispersion of UseRatio (UseRatioDisp) over the 6 repeated measurements will be measured by the intra-patient interquartile range

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital of Montpellier, Montpellier
  - Jerome FROGER, Nîmes

IPD SHARING:
Plan to Share IPD: No